CLINICAL TRIAL: NCT05968690
Title: A Phase I Study to Evaluate the Safety of Naltrexone and Propranolol in Combination With Standard of Care Ipilimumab and Nivolumab in Patients With Advanced Melanoma
Brief Title: Naltrexone and Propranolol Combined With Immunotherapy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sarah Weiss (Other)
Responsible Party: Sponsor-Investigator, Sarah Weiss, Associate Professor of Medicine, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 092302; Pro2023001214 (Other: Rutgers, The State University of New Jersey); NCI-2023-06872 (Other: NCI CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2023-07-18; First posted 2023-08-01 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Advanced Melanoma
Keywords: Melanoma; Metastatic melanoma; Skin cancer; Immune checkpoint inhibitors; Propranolol; Naltrexone; Beta-adrenergic blocker; Opioid receptor antagonist; Tumor microenvironment; NK cells; T-cells; Combination therapy; Immunotherapy; Ipilimumab; Nivolumab
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Propranolol; Naltrexone

STUDY DESIGN:
Intervention Model Description: This is an open-label, single institution, phase I study with a 3+3 design of dose escalated naltrexone in combination with propranolol 30 mg bid and ipilimumab 3 mg/kg plus nivolumab 1 mg/kg q3wk for up to 4 doses followed by NIVO monotherapy q4wk in participants with advanced melanoma.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 - Propranolol (Experimental): Patients will receive intravenous ipilimumab 3 mg/kg + nivolumab 1 mg/kg every 21 days for up to 4 cycles followed by intravenous nivolumab monotherapy 480 mg every 28 days.
  Propranolol will be administered as 30 mg orally twice a day, continuously.
  Interventions: Drug: Propranolol
- Cohort 2 - Propranolol + Naltrexone 4.5 mg (Experimental): Patients will receive intravenous ipilimumab 3 mg/kg + nivolumab 1 mg/kg every 21 days for up to 4 cycles followed by intravenous nivolumab monotherapy 480 mg every 28 days.
  Propranolol will be administered as 30 mg orally twice a day, continuously.
  Naltrexone will be administered as 4.5 mg orally once a day, continuously.
  Interventions: Drug: Propranolol; Drug: Naltrexone
- Cohort 3 - Propranolol + Naltrexone 9 mg (Experimental): Patients will receive intravenous ipilimumab 3 mg/kg + nivolumab 1 mg/kg every 21 days for up to 4 cycles followed by intravenous nivolumab monotherapy 480 mg every 28 days.
  Propranolol will be administered as 30 mg orally twice a day, continuously.
  Naltrexone will be administered as 9 mg orally once a day, continuously.
  Interventions: Drug: Propranolol; Drug: Naltrexone
- Cohort 4 - Propranolol + Naltrexone 25 mg (Experimental): Patients will receive intravenous ipilimumab 3 mg/kg + nivolumab 1 mg/kg every 21 days for up to 4 cycles followed by intravenous nivolumab monotherapy 480 mg every 28 days.
  Propranolol will be administered as 30 mg orally twice a day, continuously.
  Naltrexone will be administered as 25 mg orally once a day, continuously.
  Interventions: Drug: Propranolol; Drug: Naltrexone

INTERVENTIONS:
Drug: Propranolol — Propranolol will be administered to patients in all cohorts.
Drug: Naltrexone — Naltrexone will be administered to patients in cohorts 2, 3, and 4.
  Arms: Cohort 2 - Propranolol + Naltrexone 4.5 mg; Cohort 3 - Propranolol + Naltrexone 9 mg; Cohort 4 - Propranolol + Naltrexone 25 mg

SUMMARY:
Various forms of stress can promote cancer development and growth and negatively impact the immune system's response to tumors. Beta-adrenergic and opioid receptors co-exist in many cells including immune cells and are integral components of the body's response to stress. Pre-clinical studies have demonstrated that dual blockade of these receptors can decrease tumor growth and modulate the anti-tumor immune response. This clinical trial investigates the safety and potential therapeutic benefits of combining a beta-adrenergic blocker (propranolol) and an opioid receptor antagonist (naltrexone) with immune checkpoint inhibitors in patients with advanced melanoma.

DETAILED DESCRIPTION:
This is an open-label, single institution, phase I clinical trial to investigate the safety, tolerability, and preliminary efficacy of dose-escalated naltrexone (NTX) in combination with propranolol (PRO), ipilimumab (IPI), and nivolumab (NIVO) in patients with advanced melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older and able to understand and sign the informed consent form.
* Histologically confirmed diagnosis of unresectable stage III or stage IV melanoma.
* Candidate for standard of care therapy with ipilimumab 3 mg/kg + nivolumab 1 mg/kg.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Treatment-naïve or has received any number of prior lines of therapy. Prior targeted therapy is allowed, but small molecule inhibitors must be discontinued within two weeks before starting the study.
* Life expectancy of at least 6 months.
* Presence of at least one accessible site of disease to provide an on-study biopsy for tumor tissue. The biopsy may be waived after discussion with the Principal Investigator (PI) if it is deemed unfeasible. The site may be a target lesion as long as it will not be rendered unmeasurable by the biopsy procedure.
* Willingness to undergo tumor biopsy (if archival tumor is not available) prior to initiation of therapy and while on the study.
* Willingness to provide an archival specimen block, if available, for research purposes.
* Normal organ function, defined as:

  1. Absolute neutrophil count (ANC) >1500/mcL
  2. Platelets >100,000/mcL
  3. Hemoglobin (Hb) >9 g/dL
  4. Albumin >2.5 mg/dL
  5. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 times the upper limit of normal (ULN)
  6. Serum total bilirubin <1.5 times ULN or direct bilirubin < ULN for subjects with total bilirubin levels >1.5 times ULN.
* Female participants of childbearing potential should have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
* Female participants of childbearing potential should be willing to use a highly effective form of contraception (hormonal or intrauterine device) along with a condom in their male partner, or be surgically sterile, or abstain from heterosexual activity for a period of at least six months after the last dose of study medication.
* Male participants should agree to use an adequate method of contraception starting with the first dose of study therapy through at least six months after the last dose of study drug.
* Participants must have at least one measurable lesion at baseline by computed tomography (CT) or magnetic resonance imaging (MRI) as per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria. Tumor sites situated in a previously irradiated area or in an area subjected to other loco-regional therapy are not considered measurable unless there has been demonstrated progression in the lesion.
* Prior focal radiotherapy is allowed.

Exclusion Criteria:

* Presence of untreated brain metastases, unless discussed with the Principal Investigator (PI) and meet specific criteria for inclusion (treatment-naïve patients with brain metastases <10 mm, asymptomatic, without significant edema, hemorrhage, shift, or requirement for steroids or anti-seizure medications, and not in eloquent areas). These patients may potentially forego initial local treatment of the brain metastases and have them reassessed after consultation with the Neurosurgery and Radiation Oncology teams.
* Use of corticosteroids to control immune-related adverse events at enrollment. Participants who previously required corticosteroids for symptom control must be off steroids for at least two weeks. Low-dose steroid use (=10 mg of prednisone or equivalent) as corticosteroid replacement therapy for primary or secondary adrenal insufficiency is allowed.
* Failure to recover (i.e., Grade 1 or at baseline) from adverse events due to prior treatment.
* History of grade 3-4 neurologic or cardiac toxicity or life-threatening liver toxicity poorly responsive to steroids with prior anti-PD-1 therapy.
* Presence of leptomeningeal disease.
* Active autoimmune disease unrelated to the use of immune checkpoint inhibitors that has required systemic treatment in the past year (e.g., use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.
* Contraindications to the use of propranolol, including:

  1. Cardiogenic shock.
  2. Sinus bradycardia greater than first-degree block.
  3. Severe bronchial asthma.
  4. Known hypersensitivity to propranolol.
  5. Requirement for current use of an alternative beta-blocker.
  6. Uncontrolled diabetes.
  7. Uncontrolled depression.
  8. Unstable angina or myocardial infarction within 3 months of Day 1 Cycle 1.
* For enrollment into Cohort 2-4 ONLY: Contraindications to the use of naltrexone, including:

  1. Participants currently receiving opioid analgesics or anticipated to require opioid analgesics in the near future.
  2. Participants currently dependent on opioids, including those currently maintained on opiate agonists (e.g., methadone) or partial agonists (e.g., buprenorphine).
  3. Participants in acute opioid withdrawal.
  4. Individuals with a history of sensitivity to naltrexone.
* Pregnancy or breastfeeding. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she should inform her treating physician immediately. Breastfeeding must be discontinued if the mother is enrolled in this trial due to the potential risk for adverse events in nursing infants.
* Receipt of any other investigational agents or participation in a study of an investigational agent or use of an investigational device within four weeks of the first dose of treatment.
* Concurrent condition (including medical illness, active infection requiring treatment with intravenous antibiotics, or presence of laboratory abnormalities) or history of a prior condition that places the patient at unacceptable risk if treated with the study drug or confounds the ability to interpret data from the study.
* Concurrent, active malignancies in addition to those being studied, except for cutaneous squamous cell carcinoma or basal cell carcinoma.
* Active (non-infectious) pneumonitis.
* Hepatitis B (HBV) or Hepatitis C (HCV) acute or chronic infection.
* Receipt of a live vaccine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by Common Terminology Criteria for Adverse Events (CTCAE) v5.0 | initial 28 days of treatment and then for up to 2 years
Dose-limiting toxicity of naltrexone in combination with propranolol and ipilimumab plus nivolumab | initial 28 days of treatment
Recommended phase 2 dose of naltrexone in combination with propranolol and ipilimumab plus nivolumab | up to 2 years from start of treatment

SECONDARY OUTCOMES:
Objective Response Rate (ORR) by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | up to 2 years from start of treatment
Progression-Free Survival (PFS) | up to 2 years from start of treatment
Overall Survival (OS) | up to 2 years from start of treatment

OTHER OUTCOMES:
Exploratory objectives are to assess the impact of propranolol + naltrexone on the anti-tumor immune response through correlative biomarker studies performed on tumor and blood. | up to 2 years from start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Weiss, MD, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No